CLINICAL TRIAL: NCT01869790
Title: Development of "Fat" Bolus for Coverage of Higher Fat Meals.
Brief Title: Evaluation of Fats on Postprandial Glucose Control
Acronym: Nabucco
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Boston Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Prandial bolus coverage
Record Dates: First submitted 2013-06-02; First posted 2013-06-05 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Meal challenge (Experimental): Different fat types
  Interventions: Other: Different fat types

INTERVENTIONS:
Other: Different fat types — Saturated, monounsaturated fats

SUMMARY:
The purpose of this study is examine the effect of different fat types on postprandial glucose control in patients with type 1 diabetes.

Subjects will have several admissions and, in random order, will receive lunches with identical carbohydrate content but different fat content: lunch A will minimal fat content, lunch B will contain added butter, lunch C will contain added olive oil, and lunch D will contain added cheese. Total fat content in lunches B-D will be the same. Subjects will receive identical insulin doses (calculated using the subject's usual insulin-to-carbohydrate ratio) for the meals.

The investigators hypothesize that, despite identical carbohydrate content,the lunches higher in saturated fat will lead to more postprandial hyperglycemia than the lunch containing minimal fat and the lunch high in monounsaturated fat.

The hypothesis is that from time points 0-180 minute area under the curve for Lunches A, B, C, and D will be the same, whereas from time points 180-360 minutes for Lunch B and D will be greater than that of Lunch A and C.

DETAILED DESCRIPTION:
Subjects for this study will be adults with type 1 diabetes who use insulin pump in their diabetes self-management. Prior to admission the the clinical research center the basal rates and insulin-to-carbohydrate ratio of the subjects will be optimized using standard clinical procedures.

Subjects will be admitted to the clinical research center in mid-morning following a light breakfast at home. Subjects will have several admissions and, in random order, will receive lunches with identical carbohydrate content but different fat content: lunch A will minimal fat content, lunch B will contain added butter, lunch C will contain added olive oil, and lunch D will contain added cheese. Total fat content in lunches B-D will be the same. Subjects will receive identical insulin doses (calculated using the subject's usual insulin-to-carbohydrate ratio) for the meals. Blood samples for measurement of plasma glucose and insulin levels will be drawn for the subsequent 6 hours. We hypothesize that postprandial glucose levels 3-6 hours after start of the meal will be higher following lunches B and D, compared to lunches A and C.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18-75 years) with type 1 diabetes > 3 years.
* On insulin pump therapy.
* A1c < 8.5%.

Exclusion Criteria:

* History or symptoms suggestive of gastric dysmotility, celiac disease, pancreatic exocrine dysfunction or other conditions that cause malabsorption or maldigestion.
* Eating disorder.
* Diet allergies.
* Special diet restrictions, such as vegan or any nut allergy.
* Medications know to affect insulin sensitivity (such as glucocorticoids) or affect gastrointestinal motility (such as reglan).
* High-titre insulin autoantibodies with delayed insulin kinetics.
* Women who are breast feeding, pregnant, or wanting to become pregnant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) | 0-180 minutes vs 180-360 minutes
  One-way repeated measures ANOVA will be used to analyze area under curve differences between the three lunches as well as time in target range (80-180 mg/dL), peak blood glucose, time to peak blood glucose, time to return to baseline blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Howard Wolpert, MD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No